CLINICAL TRIAL: NCT05911386
Title: Multiparametric Echocardiography and Cardiac Biomarkers in Pediatric Inflammatory Heart Diseases (Including Pediatric Inflammatory Multisystemic Syndromes Related to Covid 19, Kawasaki Disease and Myocarditis)
Brief Title: Multiparametric Echocardiography and Cardiac Biomarkers in Pediatric Inflammatory Heart Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOSSER Gilles, chief of congenital and pediatric cardiology department, Central Hospital, Nancy, France
Other Study IDs: 2023PI058
Record Dates: First submitted 2023-05-09; First posted 2023-06-22 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Myocarditis; Pediatric Inflammatory Multisystem Syndrome; Kawasaki Disease
MeSH Terms: conditions — Myocarditis; pediatric multisystem inflammatory disease, COVID-19 related; Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MYOCARDITIS: No intervention Study of available clinical, biological, and echocardiographic data
  Interventions: Other: study of biological samples and echocardiographic data and link with need of hemodynamic support
- KAWASAKI: No intervention Study of available clinical, biological, and echocardiographic data
  Interventions: Other: study of biological samples and echocardiographic data and link with need of hemodynamic support
- PIMS: No intervention Study of available clinical, biological, and echocardiographic data
  Interventions: Other: study of biological samples and echocardiographic data and link with need of hemodynamic support

INTERVENTIONS:
Other: study of biological samples and echocardiographic data and link with need of hemodynamic support — observational study : there is no intervention

SUMMARY:
Acquired inflammatory or infectious cardiac diseases, in pediatrics, include Kawasaki disease, myocarditis, and Covid-19-related Pediatric Multisystemic Inflammatory Syndrome (PIMS).

These 3 inflammatory cardiac diseases have clinical, biological, and echographic similarities and differences. Nevertheless their modalities of monitoring, management and evolution are different. The investigators wish to retrospectively analyze biological and echocardiographic data of Kawasaki disease, myocarditis, PIMS patients managed at Nancy Children Hospital from January 1, 2017 to June 31, 2023.

The primary objective of this study is to identify, for these 3 pathologies, the prognostic factors of initiation of inotropic support.

The secondary objective is to identify the prognostic factors of degradation of ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic of PIMS, myocarditis or kawasaki disease patients
* age < 18 years

Exclusion Criteria:

* uncertain diagnosis
* other complex heart disease
* management out of Nancy University children hospital center

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: age < 18 years initial management and follow up in Nancy university children hospital center for PIMS Myocarditis and Kawasaki disease patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
need of hemodynamic support | up to 20 days
  The need for haemodynamic support is defined dichotomously: yes or no. The investigators wish to identify the predictive factors of need for haemodynamic support among the following variables: groups (PIMS, KAWASAKI, MYOCARDITIS), cardiac biomarkers (troponin and NT-pro-BNP at admission (in ng/ml)) and echocardiographic criterias (Left Ventricular Ejection fraction, global and regional longitudinal strain at admission (in %)).

SECONDARY OUTCOMES:
deterioration of Left Ventricular Ejection fraction | up to 20 days
  Left Ventricular Ejection fraction degradation is defined as an Left Ventricular Ejection fraction below the value of the first quartile of Left Ventricular Ejection fraction of all patients taken into account (Left Ventricular Ejection fraction as a percentage).
  The investigators wish to identify the predictive factors of Left Ventricular Ejection fraction degradation among the following variables: groups (PIMS, KAWASAKI, MYOCARDITIS), cardiac biomarkers (troponin and NT-pro-BNP at admission (in ng/ml)) and echocardiographic criterias (Left Ventricular Ejection fraction , global and regional longitudinal strain at admission (in %)).

CONTACTS AND LOCATIONS:
Locations (1):
- Gilles BOSSER, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No